CLINICAL TRIAL: NCT03395379
Title: Air Dissection in Percutaneous Radiofrequency Ablation of T1a Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: URO-BASE01
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Unrecognized Condition
Keywords: Radiofrequency; Thermal Protection; Percutaneous thermal ablation; Kidney neoplasms
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: RFA without air dissection protection
  Interventions: Procedure: RFA
- Group 2: RFA with air dissection protection
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: RFA — Radiofrequency ablation (RFA) is a medical procedure in which part of the electrical conduction system of the tumor is ablated using the heat generated from medium frequency alternating current.

SUMMARY:
The investigators aimed to evaluate the feasibility and safety of using ambient air to protect against thermal injury during RadioFrequency Ablation (RFA) for Renal Cell Carcinoma (RCC) based on data from cases at their institute.

DETAILED DESCRIPTION:
The incidence of renal cell carcinoma (RCC) has been increasing, particularly among patients >65 years of age. As older individuals are at higher risk for surgical complications, the use of radiofrequency ablation (RFA) for small renal masses (SRM) <4 cm in size, which include T1a tumors,may be a compelling treatment option for elderly patients. However, RFA uses heat to destroy abnormal tissue, with the risk of thermal injury to tissues and organs, including gastric tissue and nerve roots, which are in proximity to the targeted treatment zone. The incidence rate of major complication with RFA, including thermal wounds, has been reported to vary between 3.2% and 5.2%. Different thermal protection methods have been developed to lower the risk of injury to adjacent tissues during ablation, such as air dissection using CO2 injection and hydrodissection using G5% for shielding. Although both of these options are effective, they are expensive. To lower the cost of thermal protection, the investigators have been using ambient air instead of CO2 for air dissection prior to RFA for SRM-RCCs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Renal Cell Carcinoma (RCC)
* Patients with a single SRM of <4 cm, confirmed as RCC on biopsy
* RCC status : pT1a
* Eligible patients for an RadioFrequency Ablation (RFA) treatment

Exclusion Criteria:

* Patients who have already received a RFA treatment for an other tissu or tumor
* Patients who have a bleeding tumor or prior local treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study cohort is selected from our institution. Patients with a single SRM of <4 cm, confirmed as RCC on biopsy, are offered RFA as an alternative to open resection. In cases in which vital tissues are located within 10 mm of the target treatment area, air dissection are planned if the patient provide his consent.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-01-11 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-05-15 (Actual)

PRIMARY OUTCOMES:
Failure rate of the air dissection procedure | 6 weeks post-operative
  The failure rate of the air dissection procedure is defined as the need for another dissection method, the inability to create sufficient space for successful dissection and/or damage to surrounding vital tissues.

SECONDARY OUTCOMES:
Post-operative complications | 6 weeks post-operative
  Minor and major complications are recorded, corresponding to Clavien Dindo classification

IPD SHARING:
Plan to Share IPD: No
Submission at several congress: WCE2016, EAU2017, AUA2017 Publication at the Journal of Urology in December 2017

REFERENCES:
- [Background] Luciani LG, Cestari R, Tallarigo C. Incidental renal cell carcinoma-age and stage characterization and clinical implications: study of 1092 patients (1982-1997). Urology. 2000 Jul;56(1):58-62. doi: 10.1016/s0090-4295(00)00534-3. PMID 10869624
- [Background] Turrentine FE, Wang H, Simpson VB, Jones RS. Surgical risk factors, morbidity, and mortality in elderly patients. J Am Coll Surg. 2006 Dec;203(6):865-77. doi: 10.1016/j.jamcollsurg.2006.08.026. PMID 17116555
- [Background] Boss A, Clasen S, Kuczyk M, Anastasiadis A, Schmidt D, Claussen CD, Schick F, Pereira PL. Thermal damage of the genitofemoral nerve due to radiofrequency ablation of renal cell carcinoma: a potentially avoidable complication. AJR Am J Roentgenol. 2005 Dec;185(6):1627-31. doi: 10.2214/AJR.04.1946. PMID 16304025
- [Background] Joniau S, Tsivian M, Gontero P. Radiofrequency ablation for the treatment of small renal masses: safety and oncologic efficacy. Minerva Urol Nefrol. 2011 Sep;63(3):227-36. PMID 21993321
- [Background] Pieper CC, Fischer S, Strunk H, Meyer C, Thomas D, Willinek WA, Hauser S, Nadal J, Schild H, Wilhelm K. Percutaneous CT-Guided Radiofrequency Ablation of Solitary Small Renal Masses: A Single Center Experience. Rofo. 2015 Jul;187(7):577-83. doi: 10.1055/s-0034-1399340. Epub 2015 Apr 21. PMID 25962750
- [Background] Arellano RS, Garcia RG, Gervais DA, Mueller PR. Percutaneous CT-guided radiofrequency ablation of renal cell carcinoma: efficacy of organ displacement by injection of 5% dextrose in water into the retroperitoneum. AJR Am J Roentgenol. 2009 Dec;193(6):1686-90. doi: 10.2214/AJR.09.2904. PMID 19933665
- [Background] Laeseke PF, Sampson LA, Brace CL, Winter TC 3rd, Fine JP, Lee FT Jr. Unintended thermal injuries from radiofrequency ablation: protection with 5% dextrose in water. AJR Am J Roentgenol. 2006 May;186(5 Suppl):S249-54. doi: 10.2214/AJR.04.1240. PMID 16632684
- [Background] Farrell MA, Charboneau JW, Callstrom MR, Reading CC, Engen DE, Blute ML. Paranephric water instillation: a technique to prevent bowel injury during percutaneous renal radiofrequency ablation. AJR Am J Roentgenol. 2003 Nov;181(5):1315-7. doi: 10.2214/ajr.181.5.1811315. No abstract available. PMID 14573426
- [Background] Zlotta AR, Wildschutz T, Raviv G, Peny MO, van Gansbeke D, Noel JC, Schulman CC. Radiofrequency interstitial tumor ablation (RITA) is a possible new modality for treatment of renal cancer: ex vivo and in vivo experience. J Endourol. 1997 Aug;11(4):251-8. doi: 10.1089/end.1997.11.251. PMID 9376843
- See also: Recommandations en onco-urologie 2013 du CCAFU: Cancer du rein — http://preprod.oncolr.org/upload/Espace_patients/Referentiels_regionaux/RPC_CCAFU_Krein_Prog13.pdf
- See also: Thermal protection during percutaneous thermal ablation procedures: interest of carbon dioxide dissection and temperature monitoring. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4916825/
- See also: Minimizing diaphragmatic injury during radiofrequency ablation: efficacy of intra-abdominal carbon dioxide insufflation — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3834111/
- See also: Thermal protection during percutaneous thermal ablation of renal cell carcinoma. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2408950/
- See also: Thermal protection with 5% dextrose solution blanket during radiofrequency ablation. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2443416/